CLINICAL TRIAL: NCT00413777
Title: A Phase 2, Multi-center, Open-label Study to Determine Long-term Safety, Tolerability and Efficacy of Split-dose Oral Regimens of Tolvaptan Tablets in a Range of 30 to 120 mg/d in Patients With Autosomal Dominant Polycystic Kidney Disease
Brief Title: Tolvaptan Open-label Pilot Efficacy, Tolerability, and Safety Study in Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Acronym: TEMPO 2:4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 156-04-250
Record Dates: First submitted 2006-12-18; First posted 2006-12-20 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-05

CONDITIONS: Polycystic Kidney, Autosomal Dominant
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Tolvaptan

ARMS (2):
- Tolvaptan 45/15 mg/day orally for up to 4 years (Experimental): Participants received tolvaptan 45 mg orally in the morning and 15 mg orally 8 hours later for up to 4 years.
  Interventions: Drug: Tolvaptan
- Tolvaptan 60/30 mg/day orally for up to 4 years (Experimental): Participants received tolvaptan 60 mg orally in the morning and 30 mg orally 8 hours later for up to 4 years.
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — Participants were titrated to either the tolvaptan 45/15 or 60/30 mg split-dose over a 2-month Titration Period. They received the titrated dose for 34 months during the Fixed-dose Period. Following a planned off-treatment period, participants had the option to enter an Extension Period for an additional 12 months. Tolvaptan was supplied as tablets.
  Other Names: OPC-41061

SUMMARY:
This study's purpose is to evaluate the long-term safety of open-label tolvaptan regimens to determine the maximally-tolerated dose and acquire pilot efficacy data in patients with autosomal dominant polycystic kidney disease (ADPKD).

DETAILED DESCRIPTION:
Autosomal Dominant Polycystic Kidney Disease is a genetic disease classified by the formation of fluid-filled cysts in the kidneys. The accumulation of these cysts causes the kidneys to enlarge several times the normal size and leads to the eventual loss of renal function and ultimately results in renal failure in end-stage patients. This is a disease with life-threatening implications to those who have it, and their family members who may also be affected. Aside from early anti-hypertensive control and dietary protein restriction, which are presumed to offer a modest degree of protection, most surviving patients require renal replacement therapy (dialysis and transplant) and suffer from high morbidity and mortality.

A rationale for use of tolvaptan in these genetic disorders has been proven, in principle, through use of a variety of animal models. In these models, tolvaptan is effective in halting or reversing the progression of this renal disease.

The current study is being undertaken in order to evaluate whether tolvaptan, an oral vasopressin V2 receptor inhibitor, will maintain an adequate safety profile and show a potential clinical benefit by reducing total renal volume in the hopes of making an impact upon disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Prior participation in designated tolvaptan ADPKD studies (156-04-248, 156-04-249).
* Able to give Informed Consent.

Exclusion Criteria:

* Women who are breast feeding and females of childbearing potential who are not using acceptable contraceptive methods.
* In the opinion of the study investigator or sponsor may present a safety risk.
* Patients who are unlikely to adequately comply with study procedures.
* Patients who at Day 1 have an estimated glomerular filtration rate (GFR) below 30 mL/min or who anticipate renal-replacement therapy within one year of study entry.
* Patients having contraindications to magnetic resonance imaging (MRI) or gadolinium contrast will be eligible but will not be able to participate in MRI.
* Patients taking a diuretic within 1 week of enrollment or likely to need diuretic therapy prior to Month 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Torres, MD, PhD, Principal Investigator — Mayo Medical Center; Frank Czerweic, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (11):
- United States (11):
  - University of Colorado, Denver, Colorado
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Univerisity of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Davita Clinical Research, Minneapolis, Minnesota
  - Mayo Medical Center, Rochester, Minnesota
  - Rogosin Institute, New York, New York
  - Northwest Renal Clinic, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Nephrology Clinical Research Center at the University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Background] Gattone VH 2nd, Wang X, Harris PC, Torres VE. Inhibition of renal cystic disease development and progression by a vasopressin V2 receptor antagonist. Nat Med. 2003 Oct;9(10):1323-6. doi: 10.1038/nm935. Epub 2003 Sep 21. PMID 14502283
- [Background] Torres VE, Wang X, Qian Q, Somlo S, Harris PC, Gattone VH 2nd. Effective treatment of an orthologous model of autosomal dominant polycystic kidney disease. Nat Med. 2004 Apr;10(4):363-4. doi: 10.1038/nm1004. Epub 2004 Feb 29. PMID 14991049
- [Result] Higashihara E, Torres VE, Chapman AB, Grantham JJ, Bae K, Watnick TJ, Horie S, Nutahara K, Ouyang J, Krasa HB, Czerwiec FS; TEMPOFormula and 156-05-002 Study Investigators. Tolvaptan in autosomal dominant polycystic kidney disease: three years' experience. Clin J Am Soc Nephrol. 2011 Oct;6(10):2499-507. doi: 10.2215/CJN.03530411. Epub 2011 Sep 8. PMID 21903984
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Lioudis M, Zhou X, Davenport E, Nunna S, Krasa HB, Oberdhan D, Fernandes AW. Effects of tolvaptan discontinuation in patients with autosomal dominant polycystic kidney disease: a post hoc pooled analysis. BMC Nephrol. 2023 Jun 22;24(1):182. doi: 10.1186/s12882-023-03247-6. PMID 37349694
- [Derived] Chebib FT, Zhou X, Garbinsky D, Davenport E, Nunna S, Oberdhan D, Fernandes A. Tolvaptan and Kidney Function Decline in Older Individuals With Autosomal Dominant Polycystic Kidney Disease: A Pooled Analysis of Randomized Clinical Trials and Observational Studies. Kidney Med. 2023 Apr 14;5(6):100639. doi: 10.1016/j.xkme.2023.100639. eCollection 2023 Jun. PMID 37250503

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A phase 2, multi-center, open-label trial, to determine the safety, tolerability, and efficacy study of split-dose oral regimens of tolvaptan tablets in a range of 30 to 120 mg/d in autosomal dominant polycystic kidney disease (ADPKD) participants.
Pre-assignment Details: This was an open-label study with a 30-day Screening period, Titration period (Day 1 to Month 2), Fixed-dose period (Month 2 to Month 36), and Extension period (12 Months).
Groups:
- Tolvaptan 45+15 mg: Participants had received tolvaptan tablets of 45+15 mg orally twice daily during the fixed-dose period from Month 2 to Month 36 followed by a planned extension period for an additional 12 Months.
- Tolvaptan 60+30 mg: Participants had received tolvaptan tablets of 60+30 mg orally twice daily during the fixed-dose period from Month 2 to Month 36 followed by a planned extension period for an additional 12 Months.
Period: Fixed-dose Period
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Started (Screened N=47; Titration period N=46; Subjects were randomized only at Fixed dose period, as above) | 22 | 24
Completed | 18 | 21
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Met Withdrawal Criteria | 1 | 0
Not completed — Withdrew Consent | 0 | 1
Period: Extension Period
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.3 (8.4) | 43.9 (7.8) | 41.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety Assessments Based on Vital Signs, Electrocardiogram (ECG's), Clinical Laboratory Tests, Physical Examinations Are Reported as Adverse Events (AEs) Upon Study Physician Discretion.
Description: An AE was defined as any new medical problem, or exacerbation of an existing problem, experienced by a participant while enrolled in a study , whether or not it was considered drug-related by the study physician. A treatment-emergent AE (TEAE) was defined as an AE that started after start of study drug treatment; or if the event was continuous from Baseline and was serious, study drug related, or resulted in death, discontinuation.
Time Frame: AEs were recorded from screening (ICF was signed) until 7-Day follow-up
Population: Safety dataset was defined as all participants who consumed at least 1 dose of study medication. Safety variables analyzed included physical examinations, laboratory tests, vital signs, ECG's and AEs.
Measure: Number; unit: participants
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 22 | 24
participants
  Participants with serious TEAEs | 3 | 8
  Participants with severe TEAEs | 6 | 10
  Participants discontinued due to AEs | 3 | 1

2. Secondary Outcome: Mean Change From Baseline in Trough Urine Osmolality at Steady State Prior to First Daily Dose.
Description: Spot urine osmolality at trough was determined for urine samples collected immediately prior to morning dosing for Day 1 (Baseline), Months 2, 6, 12, 24, 36 for all participants. Sample was taken after the first morning's void and was provided as a mid-stream, clean catch sample. During the titration period (Weeks 1, 2, 3 and 4) and at Month 6, additional samples were collected for the preceding day immediately preceding the 2nd daily dose and at bed-time. These samples allowed derivation of an average nadir of spot urine osmolality concentrations at each dose level and while at steady state during extended tolvaptan administration. At the Month 36 visit, participants were given a urine container and brought back the specimen at Extension Day 1. All participants were fasting.
Time Frame: Baseline to Month 36
Population: The intent-to-treat (ITT) dataset was defined as a dataset that included data from all participants who enrolled to the study with observations at Baseline and Post Baseline. Observed cases (OC) dataset were used.
Measure: Mean (Standard Deviation); unit: mOsm/kg
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 22 | 24
mOsm/kg
  Month 2 (N= 21, 22) | -274.10 (223.14) | -228.00 (238.19)
  Month 6 (N= 19, 23) | -288.42 (219.55) | -263.78 (221.05)
  Month 12 (N= 17, 21) | -227.29 (226.63) | -178.43 (228.43)
  Month 24 (N= 18, 20) | -170.17 (272.21) | -189.75 (229.33)
  Month 36 (N= 18, 21) | -222.50 (229.91) | -208.90 (194.19)

3. Secondary Outcome: Mean Change From Baseline in Trough Urine Osmolality at Steady State Prior to Second Daily Dose.
Description: Urine osmolality at steady state (after at least 4 days of dosing) including "absolute trough" prior to the second daily dose.
  Samples for this assessment were taken as closely coincident to PK blood sample as practical. During Weeks 1, 2, 3 and 4 of the Titration Period and at Month 6, additional samples were collected for the preceding day immediately preceding the second daily dose. These samples allowed derivation of an average nadir of spot urine osmolality concentrations at each dose level and while at steady state during extended tolvaptan administration.
Time Frame: Baseline to Month 24
Population: The ITT dataset was defined as a dataset that included data from all participants who enrolled to the study with observations at Baseline and Post Baseline. OC dataset were used.
Measure: Mean (Standard Deviation); unit: mOsm/kg
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 20 | 24
mOsm/kg
  Month 2 (N= 21, 21) | -263.95 (220.40) | -298.71 (257.53)
  Month 6 (N= 19, 23) | -321.78 (242.53) | -294.13 (215.95)
  Month 12 (N= 16, 20) | -288.20 (216.85) | -234.65 (238.82)
  Month 24 (N= 1, 7) | -405.00 (NA) — The standard deviation value was not available or not determined. | -227.14 (334.13)

4. Secondary Outcome: Mean Change From Baseline in Trough Urine Osmolality at Steady State Prior to Bedtime.
Description: Urine osmolality at steady state (after at least 4 days of dosing) including "average of troughs" (the mean urine osmolality prior to bedtime).
  Samples for this assessment were to be taken as closely coincident to PK blood sample as practical. During Weeks 1, 2, 3 and 4 of the Titration Period and at Month 6, additional samples were collected for the preceding day at bedtime. These samples allowed derivation of an average nadir of spot urine osmolality concentrations at each dose level and while at steady state during extended tolvaptan administration.
Time Frame: Baseline to Month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mOsm/kg
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 19 | 24
mOsm/kg
  Month 2 (N= 21, 22) | -275.00 (219.37) | -291.09 (194.88)
  Month 6 (N= 19, 23) | -327.41 (217.15) | -301.83 (210.55)
  Month 12 (16, 18) | -283.21 (230.81) | -245.83 (234.46)
  Month 24 (N= 1, 7) | -263.00 (NA) — The standard deviation value was not available or not determined. | -246.00 (208.50)

5. Secondary Outcome: Percent Change From Baseline in Renal Volume.
Description: Total Kidney Volume (TKV) was assessed by the central magnetic resonance imaging (MRI) rater.
Time Frame: Baseline to Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage change per month
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 22 | 24
Percentage change per month
  Month 2 (N= 21, 24) | -1.0 (5.2) | -1.3 (5.3)
  Month 12 (N= 18, 22) | 0.3 (6.0) | 2.4 (6.6)
  Month 24 (N= 18, 21) | 4.6 (8.4) | 1.0 (8.3)
  Month 36 (N= 18, 20) | 9.9 (11.8) | 5.3 (10.0)

6. Secondary Outcome: Change From Pre-dose Baseline in Renal Function Estimated by Glomerular Filtration Rate (GFR).
Description: GFR was estimated using reciprocal serum creatinine formula. The formula does not adjust for body weight or height, but this may be done to normalize to body surface area. The formula for reciprocal Serum creatinine is: 1/Pcr. (Pcr = serum creatinine concentration [mg/dL]). Clinic weight scales were calibrated at least yearly.
Time Frame: Baseline to Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: dL/mg
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 22 | 24
dL/mg
  Month 2 (N= 22, 24) | -0.09 (0.11) | -0.05 (0.13)
  Month 6 (N= 19, 21) | -0.03 (0.10) | -0.01 (0.12)
  Month 9 (N= 18, 23) | -0.01 (0.12) | -0.03 (0.13)
  Month 12 (N= 17, 22) | -0.03 (0.11) | -0.01 (0.18)
  Month 16 (N= 18, 21) | -0.06 (0.12) | -0.02 (0.12)
  Month 20 (N= 18, 21) | -0.06 (0.10) | -0.03 (0.15)
  Month 24 (N= 18, 20) | -0.04 (0.10) | -0.02 (0.13)
  Month 28 (N= 18, 21) | -0.07 (0.10) | -0.02 (0.14)
  Month 32 (N= 18, 21) | -0.09 (0.14) | -0.06 (0.12)
  Month 36 (N= 18, 21) | -0.07 (0.11) | -0.06 (0.13)

7. Secondary Outcome: Mean Change From Baseline in Trough Urine Osmolality at Steady State Prior to First Daily Dose- Extension.
Description: Spot urine osmolality at trough was determined for urine samples collected immediately prior to morning dosing for Day 1 (Baseline), Months 2, 6, 12, 24, 36, Extension Day 1, and Extension Month 12 for all participants. Sample was taken after the first morning's void and was provided as a mid-stream, clean catch sample. During the titration period (Weeks 1, 2, 3 and 4) and at Month 6, additional samples were collected for the preceding day immediately preceding the 2nd daily dose and at bed-time. These samples allowed derivation of an average nadir of spot urine osmolality concentrations at each dose level and while at steady state during extended tolvaptan administration. At the Month 36 visit, participants were given a urine container and brought back the specimen at Extension Day 1. All participants were fasting.
Time Frame: Baseline to Months 2, 6, 12, 24, 36, Extension Day 1, Extension Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mOsm/kg
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 17 | 18
mOsm/kg
  Month 2 (N= 17, 17) | -328.06 (207.05) | -176.88 (225.54)
  Month 6 (N= 17, 18) | -270.94 (200.29) | -223.50 (211.61)
  Month 12 (N= 16, 17) | -234.56 (232.01) | -155.65 (242.53)
  Month 24 (N= 17, 17) | -164.06 (279.32) | -160.06 (196.50)
  Month 36 (N= 17, 18) | -234.71 (230.90) | -196.33 (175.23)
  Extension Day 1 (N= 17, 17) | -54.59 (236.96) | -157.18 (229.19)
  Extension Month 12 (N= 17, 18) | -115.59 (278.19) | -202.44 (227.92)

8. Secondary Outcome: Mean Change From Baseline in Trough Urine Osmolality at Steady State Prior to Second Daily Dose- Extension.
Description: as for outcome 3
Time Frame: Baseline to Month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mOsm/kg
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 16 | 18
mOsm/kg
  Month 2 (N= 17, 17) | -281.63 (235.90) | -254.82 (217.14)
  Month 6 (N= 17, 18) | -305.25 (223.90) | -261.61 (201.49)
  Month 12 (N= 16, 16) | -288.20 (216.85) | -190.69 (201.16)
  Month 24 (N= 1, 6) | -405.00 (NA) — The standard deviation value was not available or not determined. | -120.50 (196.05)

9. Secondary Outcome: Mean Change From Baseline in Trough Urine Osmolality at Steady State Prior to Bedtime- Extension.
Description: as for outcome 4
Time Frame: Baseline to Month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mOsm/kg
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 15 | 18
mOsm/kg
  Month 2 (N= 17, 17) | -322.27 (207.32) | -258.88 (174.51)
  Month 6 (N= 17, 18) | -309.73 (225.40) | -264.50 (180.12)
  Month 12 (16, 15) | -283.21 (230.81) | -206.00 (200.36)
  Month 24 (N= 1, 6) | -263.00 (NA) — The standard deviation value was not available or not determined. | -187.50 (153.04)

10. Secondary Outcome: Percent Change From Baseline in Renal Volume-Extension.
Description: TKV was assessed by the central magnetic resonance imaging (MRI) rater.
Time Frame: Baseline to Months 2, 12, 24, 36, Extension Day 1, Extension Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage change per month
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 17 | 18
Percentage change per month
  Month 2 (N= 17, 18) | -1.3 (5.4) | -1.4 (3.9)
  Month 12 (N= 17, 18) | -0.7 (4.5) | 1.9 (5.7)
  Month 24 (N= 17, 18) | 3.2 (6.0) | 0.2 (7.2)
  Month 36 (N= 17, 18) | 7.9 (8.7) | 3.8 (7.4)
  Extension Day 1 (N= 17, 18) | 14.1 (10.5) | 8.4 (7.9)
  Extension Month 12 (N= 17, 18) | 15.7 (12.7) | 10.7 (10.4)

11. Secondary Outcome: Change From Pre-dose Baseline in Renal Function Estimated by GFR- Extension.
Description: as for outcome 6
Time Frame: Baseline to Months 2, 6, 9, 12, 16, 20, 24, 28, 32, 36, Extension Day 1, Extension Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: dL/mg
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 17 | 18
dL/mg
  Month 2 (N= 17, 18) | -0.09 (0.11) | -0.04 (0.15)
  Month 6 (N= 17, 16) | -0.03 (0.11) | -0.00 (0.13)
  Month 9 (N= 16, 18) | -0.01 (0.11) | -0.01 (0.14)
  Month 12 (N= 16, 17) | -0.03 (0.12) | -0.00 (0.21)
  Month 16 (N= 17, 16) | -0.06 (0.12) | -0.01 (0.13)
  Month 20 (N= 17, 18) | -0.06 (0.10) | -0.02 (0.16)
  Month 24 (N= 17, 17) | -0.04 (0.11) | -0.02 (0.14)
  Month 28 (N= 17, 18) | -0.06 (0.10) | -0.02 (0.14)
  Month 32 (N= 17, 18) | -0.09 (0.14) | -0.05 (0.12)
  Month 36 (N= 17, 18) | -0.07 (0.11) | -0.05 (0.14)
  Extension Day 1 (N= 17, 18) | -0.04 (0.13) | -0.01 (0.17)
  Extension Month 12 (N= 17, 18) | -0.05 (0.17) | -0.04 (0.14)

12. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure (sBP) for Hypertension Assessment.
Description: The participants were seated and resting systolic and diastolic BP for each scheduled assessment was recorded. At each assessment, participants were categorized (based on repeated blood pressure measurements as being normotensive (MAP < 100 mm Hg and off therapy), high normal (sBP > 129 and or dBP > 84 mm Hg off therapy) or hypertensive (sBP >140 and/or dBP > 90 mm Hg). The mean arterial pressure (MAP) was derived from these values and were not recorded (MAP = diastolic pressure + [1/3 x pulse pressure (ie systolic - diastolic pressure)] in mm Hg).
Time Frame: Baseline to Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 22 | 24
mmHg
  Month 2 (N= 22, 24) | -3.2 (12.6) | -3.0 (15.4)
  Month 6 (N= 19, 23) | -3.6 (10.8) | -5.0 (12.4)
  Month 9 (N= 18, 23) | -4.6 (12.5) | -3.5 (12.5)
  Month 12 (N= 18, 23) | -8.0 (14.6) | -3.5 (14.2)
  Month 16 (N= 18, 23) | -6.2 (14.2) | -2.9 (12.6)
  Month 20 (N= 18, 21) | -7.9 (11.4) | -10.0 (16.4)
  Month 24 (N= 18, 21) | -2.1 (18.4) | -0.1 (14.7)
  Month 28 (N= 18, 21) | -4.7 (14.2) | -4.1 (17.1)
  Month 32 (N= 18, 21) | -7.3 (10.9) | -7.2 (14.8)
  Month 36 (N= 18, 21) | -0.2 (13.2) | -5.4 (17.6)

13. Secondary Outcome: Mean Change From Baseline in Diastolic Blood Pressure (dBP) for Hypertension Assessment.
Description: as for outcome 12
Time Frame: Baseline to Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 22 | 24
mmHg
  Month 2 (N= 22, 24) | -4.0 (11.4) | -0.2 (9.8)
  Month 6 (N= 19, 23) | -3.6 (8.2) | -2.5 (11.2)
  Month 9 (N= 18, 23) | -4.8 (8.9) | -2.8 (11.4)
  Month 12 (N= 17, 23) | -9.2 (12.6) | -1.1 (12.6)
  Month 16 (N= 18, 23) | -5.6 (11.4) | -2.3 (10.7)
  Month 20 (N= 18, 21) | -7.4 (9.8) | -5.6 (12.1)
  Month 24 (N= 18, 21) | -3.1 (11.6) | -0.1 (12.4)
  Month 28 (N= 18, 21) | -5.3 (10.6) | -2.2 (8.8)
  Month 32 (N= 18, 21) | -4.6 (11.2) | -3.0 (10.9)
  Month 36 (N= 18, 21) | -5.4 (10.0) | -4.0 (13.2)

14. Secondary Outcome: Mean Change From Baseline in Mean Arterial Pressure (MAP) for Hypertension Assessment.
Description: as for outcome 12
Time Frame: Baseline to Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 22 | 24
mmHg
  Month 2 (N= 22, 24) | -3.7 (10.5) | -1.0 (10.5)
  Month 6 (N= 19, 23) | -3.6 (7.4) | -3.3 (11.1)
  Month 9 (N= 18, 23) | -4.7 (9.2) | -3.0 (10.8)
  Month 12 (N= 18, 23) | -12.0 (18.9) | -1.8 (12.1)
  Month 16 (N= 18, 23) | -5.8 (11.0) | -2.5 (10.6)
  Month 20 (N= 18, 21) | -7.6 (9.7) | -7.0 (12.3)
  Month 24 (N= 18, 21) | -2.7 (13.0) | -0.1 (12.0)
  Month 28 (N= 18, 21) | -5.2 (11.2) | -2.7 (10.1)
  Month 32 (N= 18, 21) | -5.6 (10.0) | -4.3 (11.2)
  Month 36 (N= 18, 21) | -3.8 (9.6) | -4.4 (13.8)

15. Secondary Outcome: Mean Change From Baseline in sBP for Hypertension Assessment- Extension.
Description: as for outcome 12
Time Frame: Baseline to Months 2, 6, 9, 12, 16, 20, 24, 28, 32, 36, Extension Day 1, Extension Month 4, Extension Month 8, Extension Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 17 | 18
mmHg
  Month 2 (N= 17, 18) | -1.6 (13.0) | -2.7 (15.0)
  Month 6 (N= 17, 18) | -3.4 (11.4) | -5.6 (13.7)
  Month 9 (N= 16, 18) | -4.1 (13.2) | -4.3 (13.7)
  Month 12 (N= 17, 18) | -8.9 (14.5) | -3.3 (15.5)
  Month 16 (N= 17, 18) | -6.5 (14.5) | -1.7 (13.9)
  Month 20 (N= 17, 18) | -7.7 (11.7) | -9.3 (17.1)
  Month 24 (N= 17, 18) | -1.8 (18.9) | 1.4 (15.2)
  Month 28 (N= 17, 18) | -4.9 (14.6) | -3.4 (17.7)
  Month 32 (N= 17, 18) | -7.6 (11.1) | -6.8 (16.0)
  Month 36 (N= 17, 18) | -0.6 (13.5) | -5.4 (18.8)
  Extension Day 1 (N= 17, 18) | -4.4 (11.8) | -5.1 (14.9)
  Extension Month 4 (N= 17, 18) | -1.1 (16.1) | -8.7 (11.8)
  Extension Month 8 (N= 17, 18) | 1.8 (13.1) | -7.3 (14.8)
  Extension Month 12 (N= 17, 18) | -0.5 (13.5) | -7.1 (12.2)

16. Secondary Outcome: Mean Change From Baseline in dBP for Hypertension Assessment- Extension.
Description: as for outcome 12
Time Frame: as for outcome 15
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 17 | 18
mmHg
  Month 2 (N= 17, 18) | -5.5 (12.4) | 0.3 (9.7)
  Month 6 (N= 17, 18) | -4.5 (8.2) | -2.4 (12.6)
  Month 9 (N= 16, 18) | -5.3 (9.4) | -2.9 (11.8)
  Month 12 (N= 16, 18) | -10.1 (12.4) | -1.9 (13.0)
  Month 16 (N= 17, 18) | -6.9 (10.1) | -2.1 (12.0)
  Month 20 (N= 17, 18) | -7.5 (10.0) | -6.1 (12.1)
  Month 24 (N= 17, 18) | -3.9 (11.4) | -0.6 (12.7)
  Month 28 (N= 17, 18) | -5.6 (10.8) | -2.9 (8.4)
  Month 32 (N= 17, 18) | -5.4 (11.0) | -3.6 (11.4)
  Month 36 (N= 17, 18) | -5.7 (10.2) | -4.8 (14.0)
  Extension Day 1 (N= 17, 18) | -7.9 (7.3) | -4.0 (10.8)
  Extension Month 4 (N= 17, 18) | -6.8 (10.6) | -6.1 (10.8)
  Extension Month 8 (N= 17, 18) | -5.0 (7.9) | -6.7 (12.7)
  Extension Month 12 (N= 17, 18) | -6.0 (8.9) | -5.6 (11.7)

17. Secondary Outcome: Mean Change From Baseline in MAP for Hypertension Assessment- Extension.
Description: as for outcome 12
Time Frame: as for outcome 15
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 17 | 18
mmHg
  Month 2 (N= 17, 18) | -4.1 (11.6) | -0.6 (10.0)
  Month 6 (N= 17, 18) | -4.2 (7.7) | -3.4 (12.5)
  Month 9 (N= 16, 18) | -4.8 (9.8) | -3.4 (11.5)
  Month 12 (N= 17, 18) | -13.1 (18.9) | -2.3 (12.9)
  Month 16 (N= 17, 18) | -6.8 (10.4) | -1.9 (11.8)
  Month 20 (N= 17, 18) | -7.5 (10.0) | -7.2 (12.8)
  Month 24 (N= 17, 18) | -3.1 (13.2) | 0.1 (12.6)
  Month 28 (N= 17, 18) | -5.5 (11.4) | -2.9 (10.2)
  Month 32 (N= 17, 18) | -6.2 (10.0) | -4.6 (12.0)
  Month 36 (N= 17, 18) | -4.1 (9.8) | -5.1 (14.8)
  Extension Day 1 (N= 17, 18) | -6.8 (7.8) | -4.4 (11.0)
  Extension Month 4 (N= 17, 18) | -5.1 (10.7) | -6.9 (10.1)
  Extension Month 8 (N= 17, 18) | -2.8 (8.6) | -6.8 (12.1)
  Extension Month 12 (N= 17, 18) | -4.2 (9.3) | -6.0 (10.9)

18. Secondary Outcome: Mean Change From Baseline in Patient-assessed Renal Pain Scale.
Description: Participants were asked the question to assess the relative level of pain attributed to their kidneys. This question was, "On a scale of 0 to 10, with zero represented no pain at all and 10 represented the worst pain ever experienced, what was the worst kidney pain experienced in the last 4 months?" If the latest assessment was less than 4 months prior, the question was substituted "since your last visit" for "in the last 4 months". The same interrogator designated to this task was used throughout the study for each participant.
Time Frame: Baseline to Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 22 | 24
Units on a scale
  Month 2 (N= 22, 24) | 0.6 (3.1) | 0.0 (1.6)
  Month 6 (N= 19, 23) | 0.4 (2.8) | -0.1 (1.7)
  Month 12 (N= 18, 23) | 1.2 (3.3) | -0.1 (2.1)
  Month 24 (N= 18, 21) | 0.2 (1.6) | 1.0 (3.3)
  Month 36 (N= 18, 21) | 0.6 (2.3) | 0.5 (2.2)

19. Secondary Outcome: Mean Change From Baseline in Patient-assessed Renal Pain Scale- Extension.
Description: as for outcome 18
Time Frame: Baseline to Months 2, 6, 12, 24, 36, Extension Day 1, Extension Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 17 | 18
Units on a scale
  Month 2 (N= 17, 18) | 0.9 (2.7) | 0.3 (1.3)
  Month 6 (N=17, 18) | 0.8 (2.5) | -0.2 (1.9)
  Month 12 (N= 17, 18) | 1.2 (3.4) | -0.3 (2.0)
  Month 24 (N= 17, 18) | 0.2 (1.6) | 0.8 (3.3)
  Month 36 (N= 17, 18) | 0.6 (2.3) | 0.5 (2.4)
  Extension Day 1 (N= 17, 18) | -0.3 (0.6) | 0.8 (2.1)
  Extension Month 12 (N= 17, 18) | -0.4 (1.3) | -0.6 (2.2)

20. Secondary Outcome: Mean Change From Baseline in Abdominal Girth Measurement.
Description: The participant had a measurement of their abdominal girth recorded. The measurement will be taken with a tape measure extending around the abdomen at the level of the iliac crests laterally and the umbilicus anteriorly. The examiner should also palpate for each kidney and liver edge, noting presence or enlargement. (By definition if the kidneys are palpable they are enlarged, the liver edge may be palpable but not enlarged).
Time Frame: Baseline to Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 22 | 24
cm
  Month 2 (N= 22, 24) | 0.6 (5.0) | -2.3 (6.1)
  Month 6 (N= 18, 23) | 1.4 (6.5) | 0.5 (4.6)
  Month 12 (N= 18, 23) | 1.3 (4.7) | -2.8 (11.5)
  Month 24 (N= 17, 21) | 2.0 (7.4) | -0.6 (6.7)
  Month 36 (N= 18, 21) | 3.1 (7.2) | 0.3 (7.3)

21. Secondary Outcome: Mean Change From Baseline in Abdominal Girth Measurement- Extension.
Description: as for outcome 20
Time Frame: Baseline to Extension Day 1, Extension Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Number analyzed (Participants) | 17 | 18
cm
  Month 2 (N= 17, 18) | -0.8 (3.9) | -2.8 (7.0)
  Month 6 (N= 16, 18) | 0.3 (5.6) | 0.3 (5.1)
  Month 12 (N= 17, 18) | 1.1 (4.8) | -3.5 (12.9)
  Month 24 (N= 17, 21) | 2.0 (7.4) | -1.1 (7.1)
  Month 36 (N= 17, 18) | 2.5 (6.9) | 0.1 (7.7)
  Extension Day 1 (N= 17, 18) | 4.2 (7.2) | 2.9 (7.9)
  Extension Month 12 (N= 17, 18) | 4.6 (9.5) | 1.6 (6.1)

ADVERSE EVENTS:
Time Frame: AEs were recorded from screening (ICF was signed) until 7-days of safety follow-up. Participants with AEs in multiple system organ classes were counted only once towards the total.
Description: A SAE was any untoward medical occurrence resulted in death or was life-threatening or required inpatient hospitalization or prolonged hospitalization. An AE was an exacerbation of an existing problem or any new problem, experienced by a participant when enrolled in a trial, whether or not it was considered drug related by the study physician.
Arm/Group | Tolvaptan 45+15 mg | Tolvaptan 60+30 mg
Serious Adverse Events (participants affected / at risk) | 3/22 | 8/24
Other Adverse Events (participants affected / at risk) | 20/22 | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan 45+15 mg (N=22) | Tolvaptan 60+30 mg (N=24)
Atrial fibrillation (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 1
Polycystic liver disease (Congenital, familial and genetic disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Epiploic appendagitis (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumor benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Renal pain (Renal and urinary disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan 45+15 mg (N=22) | Tolvaptan 60+30 mg (N=24)
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Palpitations (Cardiac disorders) | 3 | 1
Dry eye (Eye disorders) | 3 | 2
Abdominal distension (Gastrointestinal disorders) | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Diarhhoea (Gastrointestinal disorders) | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Food poisoning (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Umbilical hernia (Gastrointestinal disorders) | 2 | 0
Chest pain (General disorders) | 3 | 2
Fatigue (General disorders) | 4 | 5
Oedema peripheral (General disorders) | 3 | 3
Thirst (General disorders) | 1 | 5
Bronchitis (Infections and infestations) | 3 | 2
Fungal infection (Infections and infestations) | 0 | 2
Gastroenteritis viral (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Otitis media (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 6
Urinary tract infection (Infections and infestations) | 1 | 6
Viral infection (Infections and infestations) | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 1 | 2
Incision site pain (Injury, poisoning and procedural complications) | 0 | 2
Weight increased (Investigations) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 6 | 3
Headache (Nervous system disorders) | 3 | 3
Anxiety (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 3
Haematuria (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Nocturia (Renal and urinary disorders) | 5 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 3
Polyuria (Renal and urinary disorders) | 6 | 2
Renal pain (Renal and urinary disorders) | 9 | 9
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 3 | 2
Hypotension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No